CLINICAL TRIAL: NCT00616915
Title: Does Sleep Quality Change After Switch From Wellbutrin SR to Wellbutrin XL in Patients With Major Depressive Disorder?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Roumen Milev, MD, Queen's University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSIY-219-05
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Mood Disorder
Keywords: Wellbutrin SR
MeSH Terms: conditions — Mood Disorders | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Wellbutrin SR switched to Wellbutrin XL
  Interventions: Drug: Wellbutrin XL

INTERVENTIONS:
Drug: Wellbutrin XL — Wellbutrin XL 300mg daily
  Other Names: Bupropion

SUMMARY:
Wellbutrin (bupropion) is an effective antidepressant (Thase, M 2005). It exists in instant release (IR), sustained release (SR) and extended release (XL) forms. The IR formulation was never approved for use in Canada. The XL formulation allows for once daily dosing.

Wellbutrin is both a norepinephrine and dopamine reuptake inhibitor, and as such increases the synaptic concentration of both neurotransmitters. This adds to its positive effects on cognition, apathy, tiredness and executive functioning. The increased activation may be also responsible for some of its side effects such as initial insomnia and reduced sleep efficiency, especially when taken at night.

DETAILED DESCRIPTION:
Wellbutrin SR formulation cannot be given as more than 150 mg as a single dose and higher doses are commonly required for the treatment of depression; they also have to be given at least 8 hours apart in order to avoid peak plasma concentrations and to reduce the risk of seizures (incidence of 0.1% at doses £ 300 mg). The twice a day dosing may result in complaints of insomnia and may necessitate discontinuing the medication or adding a sleep promoting agent. The benefit of once-daily dosing cannot be understated given treatment adherence is typically lower in depressed patients than their non-depressed counterparts; further, the 8 h dosing interval of bupropion SR is likely to have lower adherence compared with traditional bid dosing (i.e., morning and evening); thus, it is not difficult to imagine patients missing 30-50% of their second dose given the difficulty of recalling to take the second dose at work or school. The review of Fava et al. (2005) plots the relative PK profiles of XL and SR and notes the significantly lower bupropion concentration at bedtime, which is likely to reduce the occurrence of insomnia. Therefore, Wellbutrin XL may improve adherence by eliminating the second dose and Wellbutrin XL also avoids the high plasma drug concentrations at bedtime, as seen with bupropion SR, which are associated with insomnia. Further, the smoother pharmacokinetic profile of Wellbutrin XL may improve overall tolerability compared with Wellbutrin SR.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Patient Informed Consent;
2. Patients with Major Depressive Disorders (DSM-IV-TR - criteria used);
3. Out-patients;
4. Males or females over 18 years of age;
5. Patients currently using Wellbutrin SR.

Exclusion Criteria:

1. Bipolar Disorder patients;
2. Actively suicidal patients;
3. Schizophrenia, Schizoaffective or other Psychotic Disorder;
4. Pregnant women, as by pregnancy test at the beginning of the study;
5. Women in childbearing age, refusing to use appropriate contraception, or breastfeeding mothers;
6. Patients with known hypersensitivity to bupropion;
7. Patients with severe or unstable medical conditions, which in the opinion of the investigator would interfere with their progress or safety;
8. ECT or TMS treatments within the last three months;
9. Patients who did not respond to previous treatment with bupropion;
10. Patients with history of seizure disorder;
11. Patients with history of eating disorders (e.g. bulimia, anorexia nervosa);
12. Patients using sleep aiding medication (Benzodiazepines, barbiturates).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
This study is looking at the effect of Wellbutrin SR versus Wellbutrin XL on sleep quality | pre, 3-5days, 3-4weeks after wellbutrinXL

CONTACTS AND LOCATIONS:
Overall Officials: Roumen V. Milev, MD, Principal Investigator — Queen's University
Locations (1):
- Providence Care Mental Health Services, Kingston, Ontario, Canada